CLINICAL TRIAL: NCT05574426
Title: Efficacy of Movement Breaks in Real-World Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Canadian Institutes of Health Research (CIHR) (Other Government); McMaster University (Other)
Responsible Party: Principal Investigator, Jonathan Little, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H21-03417; 707246 (Other Grant/Funding Number: Canadian Cancer Society); POC-181042 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Exercise Snack; Movement Break; Sedentary Time; Lifestyle Exercise; Physical Activity Breaks; VILPA
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomized (1:1 allocation ratio) into Mobility or Cardiovascular movement break groups for 12-weeks. Both groups will perform 3-4 movement breaks on at least 3 days of the week.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will not be aware of group allocation and statistics performed on data with group identity blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiovascular Movement Breaks (Experimental): Participants will perform 3-4 exercise snacks (30-60s bursts of exercise) on at least 3 days of the week. The exercises prescribed in this arm will be designed to increase heart rate.
  Interventions: Behavioral: Movement Breaks
- Mobility Movement Breaks (Active Comparator): Participants will perform 3-4 mobility snacks (30-60s of mobility exercises or stretching) on at least 3 days of the week. The exercises prescribed in this arm are not designed to increase heart rate.
  Interventions: Behavioral: Movement Breaks

INTERVENTIONS:
Behavioral: Movement Breaks — Participants will be asked to perform 30-60 second movement breaks 3-4 times per day on at least 3 days per week.
  Other Names: Activity Snacks

SUMMARY:
The purpose of this study is to determine the efficacy of performing "exercise snacks" (short movement breaks throughout the day) on various measures of cardiometabolic health.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all eligible participants who have provided consent will undergo a baseline visit to assess pre-intervention basic anthropometrics, cardiorespiratory fitness, and provide a blood sample. Participants will then be randomized in a 1:1 ratio to one of two groups: 1) Mobility movement breaks (stretching or range of motion exercises); or 2) Cardiovascular movement breaks (designed to raise heart rate). Both groups will be encouraged to perform 3-4 daily movement breaks on at least 3 days of the week with support from an online platform and app that provides video instructions and reminders to complete the movement breaks. After 12 weeks, participants will be asked to return to the lab for the same testing performed at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Physically inactive (performing <150 minutes of moderate-to-vigorous intensity aerobic exercise per week, assessed by pre-screening Get Active Questionnaire);
2. Body Mass Index: 18.5-30.0 kg/m2;
3. Not currently diagnosed with or being treated for cardiometabolic disease (e.g., coronary artery disease, diabetes);
4. Not a current smoker;
5. Cleared to engage in physical activity using the Get Active Questionnaire and, if applicable, consultation with a Qualified Exercise Professional;
6. Access to a computer, tablet or smartphone for intervention delivery and tracking

Exclusion Criteria:

1. Chronic health condition preventing participation in exercise;
2. Lack of access to internet connection

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Little, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - University of British Columbia, Kelowna, British Columbia
  - McMaster University, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Babir FJ, Islam H, McCreary S, Vaz E, Falkenhain K, Cranston K, Jung M, Singer J, Sandilands R, Marcotte-Chenard A, Stamatakis E, Richards DL, Gibala MJ, Little JP. Technology-Enabled Exercise "Snacks" Are Feasible to Perform in a Real-World Setting: A Randomized Controlled Trial. Scand J Med Sci Sports. 2025 Aug;35(8):e70117. doi: 10.1111/sms.70117. PMID 40772837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Online recruitment primarily through use of third-party service.
Pre-assignment Details: 77 participants were included in the intention-to-treat analyses
Groups:
- Cardiovascular Movement Breaks: Participants were instructed to perform 3-4 exercise snacks (30-60s bursts of exercise) on at least 3 days of the week. The exercises prescribed in this arm were designed to increase heart rate.
- Mobility Movement Breaks: Participants were instructed to perform 3-4 mobility snacks (30-60s of mobility exercises or stretching) on at least 3 days of the week. The exercises prescribed in this arm were not designed to increase heart rate.
Period: Overall Study
Arm/Group | Cardiovascular Movement Breaks | Mobility Movement Breaks
Started | 38 | 39
Completed | 34 | 39
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cardiovascular Movement Breaks | Mobility Movement Breaks | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age in years
  Years | 54 (6) | 53 (7) | 54 (6)
Sex: Female, Male [Count of Participants; unit: Participants] — Biological sex assigned at birth
  Participants
    Female | 27 | 29 | 56
    Male | 11 | 10 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
VO2peak [Mean (Standard Deviation); unit: ml/kg/min] — Relative VO2peak from maximal cycle ergometer test
  ml/kg/min | 24.4 (4.3) | 24.6 (4.5) | 24.5 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cardiorespiratory Fitness at 12 Weeks
Description: Cardiorespiratory fitness will be assessed as the highest 30-s average from a laboratory-based graded VO2peak test on a cycle ergometer.
Time Frame: Baseline and Week 12
Population: Intention-to-treat
Measure: Mean (95% Confidence Interval); unit: ml/kg/min
Arm/Group | Cardiovascular Movement Breaks | Mobility Movement Breaks
Number analyzed (Participants) | 38 | 39
ml/kg/min | -0.6 [-1.4 to 0.2] | -1.0 [-1.7 to -0.3]

2. Secondary Outcome: Change From Baseline in Plasma Insulin
Description: A fasted venous blood sample will be obtained and insulin measured by commercial assay.
Time Frame: Baseline and 12 weeks
Population: Intention-to-treat
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Cardiovascular Movement Breaks | Mobility Movement Breaks
Number analyzed (Participants) | 38 | 39
percent change | -13 [-23 to -1] | -2 [-13 to 10]

3. Secondary Outcome: Change From Baseline in Plasma Glucose
Description: A fasted venous blood sample will be obtained and glucose measured by biochemical assay.
Time Frame: Baseline and 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Change From Baseline in Insulin Resistance
Description: A fasted venous blood sample will be obtained and insulin resistance estimated by homeostasis model assessment (HOMA) score
Time Frame: Baseline and 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline in Inflammatory Cytokines
Description: A fasted venous blood sample will be obtained and inflammatory cytokines measured by multiplex assay
Time Frame: Baseline and 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Change From Baseline in Body Mass
Description: Body mass will be measured by weigh scale
Time Frame: Baseline and 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Change From Baseline in Waist Circumference
Description: Waist circumference (in centimetres) will be measured using a measurement tape.
Time Frame: Baseline and 12 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Device-Measured Adherence to Movement Breaks
Description: Participants will wear accelerometers to assess adherence near the beginning and the end of the intervention.
Time Frame: Week 2 and week 11
Reporting Status: Not Posted

9. Secondary Outcome: Self-Reported Adherence to Movement Breaks
Description: Participants will be sent weekly surveys asking them to recall the total number of movement breaks performed that week.
Time Frame: Once per week for 12 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Movement Break Enjoyment Assessed by the Exercise Enjoyment Scale (EES)
Description: The EES is a validated, single-item 7-point scale to assess exercise enjoyment. Possible scores range from 1 (not at all) to 7 (extremely).
Time Frame: Immediately following each movement break for entire 12-week intervention
Reporting Status: Not Posted

11. Secondary Outcome: Rating of Perceived Exertion (RPE) Following Movement Breaks
Description: A 10 point RPE scale will be used to assess perceived exertion ranging from 0 (rest) to 10 (maximal).
Time Frame: Immediately following each movement break for entire 12-week intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Cardiovascular Movement Breaks | Mobility Movement Breaks
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/39
Other Adverse Events (participants affected / at risk) | 0/38 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT05574426/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT05574426/SAP_001.pdf